CLINICAL TRIAL: NCT04059224
Title: TraMel-WT: A Stratified Dual-stratum Open-label Two-stage Phase 2 Trial of Trametinib in Patients With Advanced Pretreated BRAFV600 Wild-type Melanoma
Brief Title: TraMel-WT: A Trial of Trametinib in Patients With Advanced Pretreated BRAFV600 Wild-type Melanoma
Acronym: TraMel-WT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Bart Neyns, Head of Medical Oncology, Universitair Ziekenhuis Brussel
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-BN-001
Record Dates: First submitted 2019-08-13; First posted 2019-08-16 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Stage IV Melanoma; Stage III Melanoma
Keywords: NRAS mutant; NRAS wild-type; BRAF V600 wild-type; Unresectable stage III melanoma; Stage IV melanoma; low-dose dabrafenib; dabrafenib; trametinib; Mekinist; Tafinlar
MeSH Terms: conditions — Melanoma | interventions — trametinib; dabrafenib

STUDY DESIGN:
Intervention Model Description: Stratified dual-stratum open-label two-stage single-center phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: advanced BRAF V600 wild-type/NRAS-mutant melanoma (Experimental): Patients will be treated with trametinib 2 mg once a day and dabrafenib 50 mg twice a day until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment.
  Interventions: Drug: Trametinib; Drug: Dabrafenib
- Arm B: advanced BRAF V600 wild-type/NRAS wild-type melanoma (Experimental): Patients will be treated with trametinib 2 mg once a day and dabrafenib 50 mg twice a day until disease progression, unacceptable treatment related toxicity or patient's refusal to continue study treatment.
  Interventions: Drug: Trametinib; Drug: Dabrafenib

INTERVENTIONS:
Drug: Trametinib — Trametinib 2 mg once a day by mouth.
  Other Names: TRA; Mekinist
Drug: Dabrafenib — Dabrafenib 50 mg twice a day by mouth. Dabrafenib can be uptitrated to 150 mg twice a day in case of dose-limiting trametinib-associated skin toxicity.
  Other Names: DAB; Tafinlar

SUMMARY:
This phase 2 trial will investigate the efficacy and safety of trametinib and dabrafenib in patients with advanced BRAF V600 (v-Raf murine sarcoma viral oncogene homolog B) wild-type melanoma (stratified according to BRAF V600 wild-type/NRAS (neuroblastoma Ras viral oncogene homolog) mutant and BRAF V600 wild-type/NRAS wild-type melanoma patients) that have been pretreated and progressed following treatment with PD-1- (programmed cell death-1) and CTLA-4-blocking (cytotoxic T-lymphocyte-associated antigen 4) immune checkpoint inhibitors. The investigators hypothesize that treatment with trametinib will result in objective antitumor activity. In order to improve the tolerability and optimize the dose intensity of trametinib, a minimal dose of dabrafenib will be added to prevent and manage trametinib-related skin toxicity.

DETAILED DESCRIPTION:
This will be a non-randomized stratified dual-arm open-label two-stage single-centre phase 2 trial.

Patients are eligible if they are diagnosed with BRAF V600 (v-Raf murine sarcoma viral oncogene homolog B) wild-type unresectable AJCC (American Joint Committee on Cancer) stage III or IV melanoma and are documented with progression of disease following treatment with a PD-1- (programmed cell death-1) and CTLA-4-blocking (cytotoxic T-lymphocyte-associated antigen 4) immune checkpoint inhibitor or who have a contraindication for treatment with immune checkpoint inhibitors.

Patients will be considered for study participation not earlier than 4 weeks after the last dosing of the prior therapy.

Patients will be stratified according to their NRAS (neuroblastoma RAS viral oncogene homolog) mutation status: arm A involves patients with advanced pretreated BRAF V600 wild-type/NRAS mutant melanoma; arm B involves patients with advanced pretreated BRAF V600 wild-type/NRAS wild-type melanoma.

All patients will be treated with trametinib 2 mg once a day and dabrafenib 50 mg twice a day. Throughout their study participation, patients will be continuously monitored for safety and evaluated for tumor response every 8 weeks or sooner if there is clinical suspicion of progressive disease. Patients will be treated until progression of disease, unacceptable toxicity or withdrawal of consent.

The primary endpoint of the study is the objective response rate. Secondary endpoints are progression-free survival, overall survival and safety.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* Signed written informed consent.
* Histologically confirmed advanced melanoma that is either stage III (unresectable) or stage IV (metastatic).
* Absence of a BRAF V600 mutation as determined by a validated test.
* In case of mucosal or acral melanoma, absence of a cKIT (proto-oncogene c-Kit) mutation as determined by a validated test.
* Presence of archival melanoma tissue of possibility of new biopsy for mutational testing.
* Subjects must have failed at least one prior systemic treatment with immune checkpoint inhibitors: CTLA-4 (cytotoxic T-lymphocyt antigen 4) blocking immune checkpoint inhibitors (ipilimumab or other experimental anti-CTLA-4 antibodies), PD-1 (programmed cell death 1) blocking immune checkpoint inhibitors (pembrolizumab, nivolumab or other experimental anti-PD-1 antibodies) and/or PD-L1 (programmed cell death ligand 1) blocking immune checkpoint inhibitors (avelumab, atezolizumab, durvalumab or other experimental anti-PD-L1 antibodies). Progression of disease per Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1, or per immune related response criteria (irRC) must have been documented during this treatment. Patients who are not able to undergo such treatment are also eligible.
* The presence of at least one measurable lesion per RECIST, version 1.1
* Interval between the date of the last administration of prior therapy for melanoma and the date of recruitment: a. ≥12 weeks following the date of the first administration and ≥4 weeks following the date of the last administration of CTLA-4, PD-1 or PD-L1 blocking immune checkpoint inhibitor; b. ≥4 weeks following the date of the last administration of chemotherapy (≥ 6 weeks in case of a nitrosurea or mitomycin C containing regimen); c. ≥4 weeks following major surgery or extensive radiotherapy.
* All prior anti-cancer treatment-related toxicities (except alopecia) must be ≤ grade 1 according to the Common Terminology Criteria for Adverse Events version 4 (CTCAE version 4.03; National Cancer Institute [NCI] 2010) at the time of recruitment.
* Able to swallow and retain oral medication and must not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels.
* Women of childbearing potential must have a negative serum pregnancy test within 14 days prior to recruitment and agree to use effective contraception throughout the treatment period, and for 16 weeks after the last dose of study treatment.
* Men with a female partner of childbearing potential must have either had a prior vasectomy or agree to use effective contraception from 14 days prior to administration of the first dose of study treatment, throughout the treatment period, and for 16 weeks after the last dose of study treatment.
* An Eastern Cooperative Oncology Group (ECOG) performance status
* Adequate baseline organ function as defined as follows: Absolute neutrophil count: ≥ 1.2 x 103/mm3; Hemoglobin: ≥ 9.0 g/dL; Platelet count: ≥ 75 x 103/mm3; prothrombin time/international normalized ratio and activated partial thromboplastin time: ≤ 1.5 x ULN (upper limit of normal); Albumin: ≥ 2.5 g/dL; Total bilirubin: ≤ 1.5 x ULN; aspartate aminotransferase and alanine aminotransferase: ≤ 2.5 x ULN; Calculated creatinine clearance: ≥ 50 mL/min (by use of the Cockroft-Gault formula); LVEF (left ventricular ejection fraction) ≥ LLN (lower limit of normal) by transthoracic echocardiogram

Exclusion Criteria:

* Subjects with uveal melanoma.
* Prior treatment with MAPK-pathway inhibitors
* Subjects with clinically active brain metastases (lesions should be stable and have been definitely treated with stereotactic radiation therapy, surgery or gamma knife therapy with no evidence of disease progression prior to enrollment.
* Any contra-indication for evaluation by whole body 18FDG-PET/CT (18-fluorodeoxyglucose positron emission tomography/computed tomography) and MRI (magnetic resonance imaging) of the brain.
* History of another malignancy. Exception: subjects who have been disease-free for 3 years, (i.e. subjects with second malignancies that are indolent or definitively treated at least 3 years ago) or subjects with a history of completely resected non-melanoma skin cancer.
* Current use of any prohibited medication.
* Taken an investigational drug within 28 days or 5 half-lives (minimum 14 days), whichever is shorter, prior to recruitment.
* Any serious or unstable pre-existing medical conditions (aside from malignancy exceptions specified above), psychiatric disorders, or other conditions that could interfere with the subject's safety, obtaining informed consent, or compliance with study procedures.
* Known Human Immunodeficiency Virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV) infection (subjects with laboratory evidence of cleared HBV and HCV infection will be permitted).
* No enzyme inducing anticonvulsants for ≥4 weeks prior to recruitment
* A history or evidence of cardiovascular risk including any of the following:

  a. Current LVEF < LLN; b. A QT interval corrected (QTc) for heart rate using the Bazett's formula (QTcB) ≥ 480 milliseconds; c. A history or evidence of current clinically significant uncontrolled arrhythmias. Exception: subjects with atrial fibrillation controlled for > 30 days prior to recruitment are eligible. d. A history (within 6 months prior to recruitment) of acute coronary syndromes (including myocardial infarction or unstable angina), or coronary angioplasty; e. A history or evidence of current ≥ Class II congestive heart failure as defined by the New York Heart Association (NYHA) guidelines; f. Treatment refractory hypertension defined as a blood pressure of systolic >140 mmHg and/or diastolic > 90 mm Hg which cannot be controlled by antihypertensive therapy; g. Patients with intra-cardiac defibrillators or permanent pacemakers; h. Known cardiac metastases; i. Abnormal cardiac valve morphology (≥ grade 2) documented by echocardiogram (subjects with grade 1 abnormalities [i.e., mild regurgitation/stenosis] can be entered on study). Subjects with moderate valvular thickening should not be entered on study.
* Uncorrectable electrolyte abnormalities (e.g. hypokalemia, hypomagnesemia, hypocalcemia), long QT syndrome or taking medicinal products known to prolong the QT interval.
* A history or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) including: a. Presence of predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, uncontrolled diabetes mellitus, or a history of hyperviscosity or hypercoagulability syndromes); or b. Visible retinal pathology as assessed by ophthalmic examination that is considered a risk factor for RVO or CSR such as: i. Evidence of new optic disc cupping; ii. Evidence of new visual field defects on automated perimetry; iii. Intraocular pressure >21 mmHg as measured by tonography.
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs chemically related to the study treatments, their excipients, and/or dimethyl sulfoxide (DMSO).
* Females who are nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Arm A: objective response rate on trametinib and dabrafenib | 2 years
  Objective response rate (ORR; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).
Arm B: objective response rate on trametinib and dabrafenib | 2 years
  Objective response rate (ORR; defined as the percentage of subjects with a confirmed complete response [CR] or partial response [PR] at any time per Response Evaluation Criteria in Solid Tumors [RECIST], version 1.1 [Eisenhauer 2009]).

SECONDARY OUTCOMES:
Arm A: progression-free survival on trametinib and dabrafenib | 2 years
  Progression-free survival (PFS; defined as the time from treatment initiation until the earliest date of disease progression or death due to any cause)
Arm A: overall survival on trametinib and dabrafenib | 2 years
  Overall survival (OS; defined as the time from treatment initiation until the date of death due to any cause).
Arm B: progression-free survival on trametinib and dabrafenib | 2 years
  Progression-free survival (PFS; defined as the time from treatment initiation until the earliest date of disease progression or death due to any cause)
Arm B: overall survival on trametinib and dabrafenib | 2 years
  Overall survival (OS; defined as the time from treatment initiation until the date of death due to any cause).
Arms A and B: incidence of adverse events on trametinib and dabrafenib | 2 years
  Adverse events graded by the Common Terminology Criteria of Adverse Events version 4 (CTCAE v4)

CONTACTS AND LOCATIONS:
Overall Officials: Bart Neyns, MD, PhD, Principal Investigator — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dummer R, Schadendorf D, Ascierto PA, Arance A, Dutriaux C, Di Giacomo AM, Rutkowski P, Del Vecchio M, Gutzmer R, Mandala M, Thomas L, Demidov L, Garbe C, Hogg D, Liszkay G, Queirolo P, Wasserman E, Ford J, Weill M, Sirulnik LA, Jehl V, Bozon V, Long GV, Flaherty K. Binimetinib versus dacarbazine in patients with advanced NRAS-mutant melanoma (NEMO): a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Apr;18(4):435-445. doi: 10.1016/S1470-2045(17)30180-8. Epub 2017 Mar 9. PMID 28284557
- [Background] Ranzani M, Alifrangis C, Perna D, Dutton-Regester K, Pritchard A, Wong K, Rashid M, Robles-Espinoza CD, Hayward NK, McDermott U, Garnett M, Adams DJ. BRAF/NRAS wild-type melanoma, NF1 status and sensitivity to trametinib. Pigment Cell Melanoma Res. 2015 Jan;28(1):117-9. doi: 10.1111/pcmr.12316. Epub 2014 Oct 13. No abstract available. PMID 25243813
- [Background] Long GV, Stroyakovskiy D, Gogas H, Levchenko E, de Braud F, Larkin J, Garbe C, Jouary T, Hauschild A, Grob JJ, Chiarion-Sileni V, Lebbe C, Mandala M, Millward M, Arance A, Bondarenko I, Haanen JB, Hansson J, Utikal J, Ferraresi V, Kovalenko N, Mohr P, Probachai V, Schadendorf D, Nathan P, Robert C, Ribas A, DeMarini DJ, Irani JG, Swann S, Legos JJ, Jin F, Mookerjee B, Flaherty K. Dabrafenib and trametinib versus dabrafenib and placebo for Val600 BRAF-mutant melanoma: a multicentre, double-blind, phase 3 randomised controlled trial. Lancet. 2015 Aug 1;386(9992):444-51. doi: 10.1016/S0140-6736(15)60898-4. Epub 2015 May 31. PMID 26037941